CLINICAL TRIAL: NCT05623475
Title: Evaluating the Effects of Implementing a Scenario-based Education Initiative and OSCE for Recognition and Management of Delirium: a Cluster Randomized Controlled Trial
Brief Title: Effects of Scenario-based Education Initiative and OSCE for Recognition and Management of Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: N20210318
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2022-10

CONDITIONS: Delirium
Keywords: Intensive Care Unit Syndrome; Delirium; OSCE
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 1. face-to-face delirium care session (30 minutes in duration);
  2. online learning delirium care activities (20 minutes in duration); and
  3. delirium care OSCE and reflective activity (30 minutes in duration).
  Interventions: Behavioral: OSCEs; Behavioral: Lecture; Behavioral: E-learning
- control group (Active Comparator): 1. face-to-face delirium care session (30 minutes in duration);
  2. online learning delirium care activities (20 minutes in duration)
  Interventions: Behavioral: Lecture; Behavioral: E-learning

INTERVENTIONS:
Behavioral: OSCEs — Scenario-based education intervention, including objective structured clinical examinations (OSCEs)
  Arms: experimental group
Behavioral: Lecture — Face-to-face Education using Delirium Care Flip Chart
Behavioral: E-learning — Delirium care video

SUMMARY:
Delirium is a disturbance in consciousness with reduced ability to focus, sustain, or shift attention that occurs over a short period of time and tends to fluctuate over the course of the day. 50% to 81.7% had delirium during their ICU hospitalization. Delirium is associated with increased physical restraint, ventilation use, length of ICU stay, and mortality. However, there is no established delirium care pathway in target hospital. Chen et al. (2014) demonstrated that structured assessment stations with immediate feedback may improve overall learning efficiency over an EBP workshop alone. However, no published delirium care education study has used OSCEs as an intervention for healthcare professionals. The aim is to evaluate the effects of implementing a Scenario- based education intervention, including objective structured clinical examinations (OSCEs) on delirium care among healthcare professionals. This is a knowledge translation research, builds on eight years of delirium care research in University of Wollongong, Australia. The research will be undertaken at ICUs in a medical center in northern of Taiwan. There are two phases: (1) systematic review to identify delirium screen tool, and (2) a randomized controlled trial was conducted to determine the effects of implementing a Scenario-based education intervention, including OSCE (experimental group), and on-line education only (control group) focused on recognition and management of delirium. The hypothesis is: Scenario-based education intervention, including OSCE can increase the competence and self-efficacy among healthcare professionals in delirium care.

DETAILED DESCRIPTION:
OSCEs are an integral aspect of all levels of medical education but limited to undergraduate nursing and allied health education. OSCEs are rarely used in the workplace as learning activities with nursing and allied health clinicians. This is the reason why this education initiative was innovative. OSCEs are simulated 'real life' clinical scenarios presented to clinicians who are required to demonstrate to an assessor the clinical tasks which form an OSCE scenario.

ELIGIBILITY:
Inclusion Criteria:

1. Registered nurse worked in acute care unit and care with critical patients
2. Licensed physician which undertake the post graduate year program worked in acute care unit and care with critical patients

Exclusion Criteria:

1.Unwilling to involved the research

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kee-Hsin Chen, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: 1. face-to-face delirium care session (30 minutes in duration);
  2. online learning delirium care activities (20 minutes in duration); and
  3. delirium care OSCE and reflective activity (30 minutes in duration).
  OSCEs: Scenario-based education intervention, including objective structured clinical examinations (OSCEs)
  Lecture: Face-to-face Education using Delirium Care Flip Chart
  E-learning: Delirium care video
- Control Group: 1. face-to-face delirium care session (30 minutes in duration);
  2. online learning delirium care activities (20 minutes in duration)
  Lecture: Face-to-face Education using Delirium Care Flip Chart
  E-learning: Delirium care video
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 61 | 39
Completed | 59 | 38
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 59 | 38 | 97
Age, Customized [Count of Participants; unit: Participants]
  20-24 year-old | 16 | 9 | 25
  25-34 year-old | 39 | 25 | 64
  35-44 year-old | 3 | 2 | 5
  45-54 year-old | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 37 | 92
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 59 | 38 | 97
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  Associate Degree | 9 | 5 | 14
  Bachelor Degree | 49 | 32 | 81
  Master Degree | 1 | 1 | 2
ICU training [Count of Participants; unit: Participants]
  Yes | 51 | 34 | 85
  No | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Delirium Knowledge
Description: 1. The "ICU Delirium Care Knowledge Quiz" (Traditional Chinese version ) developed by Ho et al. (2021) was used in this study.
  2. The "ICU Delirium Care Knowledge Quiz" (Traditional Chinese version ) consists of 16 multiple-choice questions, with 1 point awarded for each correct answer, and a maximum score of 16 points. The total score of the participants is analyzed as a continuous variable. The total range from 0 to 16 (minimum score: 0 point; and maximum score 16 points). Higher points represent better ICU Delirium Care Knowledge.
  3. The overall KR-20 coefficient of the questionnaire is 0.85, the intra-class correlation coefficient over a 30-day interval is 0.97, the content validity index (CVI) is 83%, and the exploratory factor analysis (EFA) demonstrates appropriate structural validity, with four factors explaining 60.87% of the total variance, indicating good reliability and validity.
Time Frame: T0(Baseline), T1(Immediately after the intervention), T2(Six weeks after the intervention)
Measure: Mean (Standard Deviation); unit: point
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 59 | 38
point
  T0 | 12.40 (1.72) | 13.26 (1.50)
  T1 | 13.08 (1.69) | 12.71 (2.02)
  T2 | 13.10 (1.81) | 13.78 (1.33)

ADVERSE EVENTS:
Time Frame: 6months
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/38
Other Adverse Events (participants affected / at risk) | 0/59 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT05623475/Prot_SAP_000.pdf